CLINICAL TRIAL: NCT06570486
Title: Contrast Between Traditional Regression Model and AI in Predicting Prolonged Stay Stay After Head and Neck Tumors
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2024-403-01
Record Dates: First submitted 2024-07-23; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- training group: For training models
- test group: Used to validate the model
- Prospective cohort: For the prospective validation of the model

SUMMARY:
This experiment is an observational study of cohort. By establishing a cohort of patients with head and neck tumors transferred to ICU after surgery, investigators compared the prediction effect of AI and the traditional prediction model on whether patients can be transferred to ICU within 24 hours of head and neck tumors. First retrospective analysis of patients after head and neck tumor surgery, medical records were collected, the test results are divided into training group and validation group according to 7:3, divided into 2 groups according to the patient ICU stay time is greater than 24 hours, the prediction model after the ICU duration of head and neck tumor surgery after more than 24 hours. At the same time, clean the data, train the AI with the data, and compare the effectiveness of both sides with the ROC. After the establishment of prediction model and AI training, the patients included in the cohort were evaluated by prediction model and AI immediately after being transferred to the ICU, predicting the possibility of transferring out of the ICU within 24 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Patients after head and neck tumors;
2. older than 18 years.

Exclusion Criteria:

1. Patients transferred to ICU twice after head and neck tumors;
2. Patients with unplanned transfer to the ICU.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Head and neck tumor postoperative patient transferred to icu
Sampling Method: Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
roll-out icu | From the date of ICU admission until the date of ICU discharge or death, whichever occurs first, assessed up to 30 days
  The time of patient transfer from ICU to the general ward was set as transfer out

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
If others need it, they can apply to us for the data, and we will provide it.

DOCUMENTS (2):
  • Study Protocol (2024-03-21): https://cdn.clinicaltrials.gov/large-docs/86/NCT06570486/Prot_000.pdf
  • Informed Consent Form (2024-03-21): https://cdn.clinicaltrials.gov/large-docs/86/NCT06570486/ICF_001.pdf